CLINICAL TRIAL: NCT07329478
Title: Effects of Muscle Specific as Compared to Movement Specific Muscle Energy Technique on Isometric Muscle Strength and Muscular Endurance in Individuals With Mechanical Neck Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUI/CTR/2025/25
Record Dates: First submitted 2025-12-29; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Neck Pain
Keywords: muscle strength; Movement Specific Muscle Energy Technique; Muscle Specific Muscle Energy Technique
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: assessor will be blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A:Muscle specific muscle energy technique (Experimental): Group A receives Muscle specific muscle energy technique. Tens and Hotpack 10 mins preceding every session.
  Interventions: Procedure: Muscle specific muscle energy technique
- B: Movement specific muscle energy technique (Experimental): Group B receives Movement specific muscle energy technique. Tens and Hotpack preceding every session for 10 mins.
  Interventions: Procedure: Movement specific muscle energy technique

INTERVENTIONS:
Procedure: Movement specific muscle energy technique — In the movement-specific group, participants received Post-Isometric Relaxation MET targeting cervical spine movements (flexion, extension, rotation, lateral flexion). For example, during right rotation:
  Active Contraction: The participant rotated left (opposite direction) with 30-50% effort against the therapist's resistance for 7-10 seconds.
  Relaxation: The participant relaxed completely. Stretching: The therapist gently moved the head towards the restricted range (right rotation) and held the stretch for 10-60 seconds.
  This technique enhances mobility and reduces muscular tension by combining contraction, relaxation, and stretching.
  Arms: B: Movement specific muscle energy technique
Procedure: Muscle specific muscle energy technique — In the muscle specific MET group, the participants were given post-isometric relaxation MET targeted at muscles of the neck region that are prone to get short, including anterior, middle and posterior Scalene, Sternocleidomastoid, Levator Scapulae and upper fibers of Trapezius muscle.
  Active Contraction: The participant rotated left (opposite direction) with 30-50% effort against the therapist's resistance for 7-10 seconds. Relaxation: The participant relaxed completely. Stretching: The therapist gently moved the head towards the restricted range (right rotation) and held the stretch for 10-60 seconds. This technique enhances mobility and reduces muscular tension by combining. Tens and Hot pack therapy for both groups preceding every session for 10 mins.
  Arms: A:Muscle specific muscle energy technique

SUMMARY:
Neck pain, prevalent in young adults due to poor posture, sedentary habits, and muscle imbalance. This study aims to compare the effects of muscle-specific versus movement-specific MET on pain, isometric muscle strength, and endurance of neck flexors and extensors. Pre- and post-intervention assessments using VAS, Modified Sphygmomanometer Dynamometer, and cranio-cervical flexion/extension tests will evaluate treatment outcomes.

DETAILED DESCRIPTION:
Neck pain, affecting nearly 75.7% of young adults, is commonly linked to poor posture, sedentary lifestyles, and muscle imbalances. If left untreated, it may lead to disability and degenerative changes. Among rehabilitation approaches, muscle energy techniques (METs) have shown effectiveness in improving pain, mobility, and function by targeting neuromuscular dysfunction. This study aims to compare the effects of muscle- specific MET with movement-specific MET on pain, isometric muscle strength, and muscular endurance of neck flexors and extensors in individuals with neck pain. A randomized control trial will be conducted using purposive sampling. Thirty participants will be divided into two groups: Group A (movement-specific MET) and Group B (muscle-specific MET), with both groups following a standard protocol of Tens and Hotpack applied for 10 mins proceeding every session for five sessions.

ELIGIBILITY:
Inclusion criteria

* Age 19-44 years.
* Both Genders (Male and Female).
* Limitation on cervical motion
* Pain ranging from 40-80 mm on visual analogue scale (VAS)

Exclusion criteria

* Participants with a positive history of fracture, surgery or trauma in the neck region, thoracic outlet syndrome, infection, any malignancy.
* Vascular syndromes such as vertebrobasilar insufficiency.
* Inflammatory, or rheumatic disorders, cervical radiculopathy, myelopathy, spondylosis, or syringomyelia.

Ages: 19 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 5 days
  Visual Analog Scale will be used for measuring pain intensity, 0 is no pain and 10 is worst pain.
Isometric muscle strength | 5 days
  Modified Sphygmomanometer Dynamometer will be used to measure isometric muscle strength. In which Higher pressure is stronger muscles; lower values suggest weakness or dysfunction.
Muscle endurance | 5 days
  Cranio-cervical flexion Test/ Cranio-cervical extension Test will be used for measuring muscle endurance. Strong contraction means normal; weakness suggests flexors/extensors' dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University Islamabad, Islamabad, Punjab Province, Pakistan